CLINICAL TRIAL: NCT02959840
Title: Is Intra-operative Acupuncture Point P6 Stimulation as Effective as Traditional Pharmacotherapy in Reducing Nausea and Vomiting During Cesarean Section With Regional Anesthesia?
Brief Title: Acupuncture Point P6 Stimulation for Reduction of Nausea and Vomiting During Cesarean
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Shaul Cohen, M.D., Director of Obstetric Anesthesia, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro20140000517
Record Dates: First submitted 2016-10-10; First posted 2016-11-09 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Nausea; Vomiting; Satisfaction
MeSH Terms: conditions — Nausea; Vomiting; Personal Satisfaction | interventions — Metoclopramide; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): No anti-emetic medications and no acupuncture point P6 stimulation prior to administration of the standardized regional anesthesia
- Metoclopramide, Ondansetron (Active Comparator): 10 mg Metoclopramide IV and 8 mg of Ondansetron IV immediately prior to administration of the standardized regional anesthesia
  Interventions: Drug: Metoclopramide; Drug: Ondansetron
- Acupressure Point P6 stimulator (Experimental): Acupuncture point P6 stimulation. This is a stimulation of the chi channel at the master of the heart (MH8 position) at the small depression of the volar surface of the distal right forearm just above the crest of the wrist. The device will be put on the patients in the operating room prior to administration of the regional anesthesia and will be removed after the cesarean section is complete.
  Interventions: Device: Acupressure Point P6 stimulator

INTERVENTIONS:
Device: Acupressure Point P6 stimulator — This device stimulates the chi channel at the master of the heart (MH8 position) at the small depression of the volar surface of the distal right forearm just above the crest of the wrist. The device is placed on patients in the operating room prior to administration of the regional anesthesia and will be removed after the cesarean section is complete. The device is removed from the patient in the operating room, before the patient is transported to the recovery room. Patients receive continuous stimulation at a level that is comfortable for the patient prior to administration of the standardized regional anesthesia.
  Arms: Acupressure Point P6 stimulator
Drug: Metoclopramide — 10 mg Reglan IV immediately prior to administration of the standardized regional anesthesia.
  Other Names: Reglan
  Arms: Metoclopramide, Ondansetron
Drug: Ondansetron — 8 mg of Zofran IV immediately prior to administration of the standardized regional anesthesia.
  Other Names: Zofran
  Arms: Metoclopramide, Ondansetron

SUMMARY:
The purpose of this study is to compare the effectiveness of acupressure point P6 stimulation versus intravenous ondansetron plus metoclopramide versus no antiemetic prophylaxis during elective cesarean section under regional anesthesia.

DETAILED DESCRIPTION:
The design of the study consists of the randomization of subjects undergoing cesarean section with regional anesthesia in one of three groups. The study is not blinded; as the participants will know which method they are being treated with because of the difference in site and nature of the acupuncture point P6 stimulation. The randomization of patients will be done by a computer to avoid bias before the informed consent form (ICF) is signed by the patients. The computer will generate three sets of random numbers for the three groups. Once the consent form is signed, the investigator will allocate the patients serially to the groups having those numbers . The randomization will be created before the study begins and will assign 180 subjects into one of the three groups to receive the treatment as follows:

Group I (n=60): Will be the control group patients and will not be given traditional medical therapy nor will receive acupuncture point P6 stimulation prior to administration of the standardized epidural anesthesia, as outlined below.

Group II (n=60): Will receive traditional medical management, consisting of 10 mg metoclopramide IV and 8 mg of ondansetron IV immediately prior to administration of the standardized regional anesthesia, as outlined below.

Group III (n=60): Will receive acupuncture point P6 stimulation. This is a stimulation of the chi channel at the master of the heart (MH8 position) at the small depression of the volar surface of the distal right forearm just above the crest of the wrist. The device will be put on the patients in the operating room prior to administration of the regional anesthesia and will be removed after the cesarean section is complete. The device will be removed from the patient in the operating room, before the patient is transported to the recovery room. Patients will receive continuous stimulation at a level that is comfortable for the patient prior to administration of the standardized regional anesthesia, as outlined below.

After the subjects have been randomly assigned to one of the three groups, subjects will receive the standardized regional anesthesia consisting of 2 milliliters (10 milligrams) of 0.5% bupivicaine and 20 micrograms of fentanyl and 100 micrograms of epinephrine. Patients will offer their subjective assessments of the level of nausea on a scale of 0-10 (0 = no nausea, 10 = worst nausea every experienced).

An Apfel score, which is used to predict the risk of experiencing post-operative nausea and vomiting (PONV), will also be determined with each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects ages 18 to 45
2. Subjects with American Society of Anesthesiologists (ASA) Class I or II
3. Subjects with elective primary or repeat cesarean delivery
4. Subjects who receive combined spinal epidural anesthesia
5. English and non-English speaking subjects will be included in the study

Exclusion Criteria:

1. Female subjects <18 years of age
2. Subjects requiring emergent cesarean delivery
3. History of placenta accrete
4. Multiple gestation pregnancy
5. ASA status III or higher
6. Current history of pregnancy induced hypertension, pre-eclampsia, or eclampsia
7. History of any chronic medication use (other than prenatal vitamins), including inhaler medications
8. Current urinary tract infection, pneumonia, or otitis media

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaul Cohen, MD, Principal Investigator — Robert Wood Johnson University Hospital
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afolabi BB, Lesi FE. Regional versus general anaesthesia for caesarean section. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD004350. doi: 10.1002/14651858.CD004350.pub3. PMID 23076903
- [Background] Arnberger M, Stadelmann K, Alischer P, Ponert R, Melber A, Greif R. Monitoring of neuromuscular blockade at the P6 acupuncture point reduces the incidence of postoperative nausea and vomiting. Anesthesiology. 2007 Dec;107(6):903-8. doi: 10.1097/01.anes.0000290617.98058.d9. PMID 18043058
- [Background] Chen HM, Chang FY, Hsu CT. Effect of acupressure on nausea, vomiting, anxiety and pain among post-cesarean section women in Taiwan. Kaohsiung J Med Sci. 2005 Aug;21(8):341-50. doi: 10.1016/S1607-551X(09)70132-9. PMID 16158876
- [Background] Duggal KN, Douglas MJ, Peteru EA, Merrick PM. Acupressure for intrathecal narcotic-induced nausea and vomiting after caesarean section. Int J Obstet Anesth. 1998 Oct;7(4):231-6. doi: 10.1016/s0959-289x(98)80044-7. PMID 15321185
- [Background] Fan CF, Tanhui E, Joshi S, Trivedi S, Hong Y, Shevde K. Acupressure treatment for prevention of postoperative nausea and vomiting. Anesth Analg. 1997 Apr;84(4):821-5. doi: 10.1097/00000539-199704000-00023. PMID 9085965
- [Background] Gan TJ, Jiao KR, Zenn M, Georgiade G. A randomized controlled comparison of electro-acupoint stimulation or ondansetron versus placebo for the prevention of postoperative nausea and vomiting. Anesth Analg. 2004 Oct;99(4):1070-1075. doi: 10.1213/01.ANE.0000130355.91214.9E. PMID 15385352
- [Background] Golembiewski J, Chernin E, Chopra T. Prevention and treatment of postoperative nausea and vomiting. Am J Health Syst Pharm. 2005 Jun 15;62(12):1247-60; quiz 1261-2. doi: 10.1093/ajhp/62.12.1247. PMID 15947124
- [Background] Habib AS, Itchon-Ramos N, Phillips-Bute BG, Gan TJ; Duke Women's Anesthesia (DWA) Research Group. Transcutaneous acupoint electrical stimulation with the ReliefBand for the prevention of nausea and vomiting during and after cesarean delivery under spinal anesthesia. Anesth Analg. 2006 Feb;102(2):581-4. doi: 10.1213/01.ane.0000189217.19600.5c. PMID 16428565
- [Background] Harmon D, Ryan M, Kelly A, Bowen M. Acupressure and prevention of nausea and vomiting during and after spinal anaesthesia for caesarean section. Br J Anaesth. 2000 Apr;84(4):463-7. doi: 10.1093/oxfordjournals.bja.a013471. PMID 10823097
- [Background] Ho CM, Hseu SS, Tsai SK, Lee TY. Effect of P-6 acupressure on prevention of nausea and vomiting after epidural morphine for post-cesarean section pain relief. Acta Anaesthesiol Scand. 1996 Mar;40(3):372-5. doi: 10.1111/j.1399-6576.1996.tb04448.x. PMID 8721471
- [Background] Ho CM, Tsai HJ, Chan KH, Tsai SK. P6 acupressure does not prevent emesis during spinal anesthesia for cesarean delivery. Anesth Analg. 2006 Mar;102(3):900-3. doi: 10.1213/01.ane.0000195553.82409.00. PMID 16492848
- [Background] Lewis IH, Pryn SJ, Reynolds PI, Pandit UA, Wilton NC. Effect of P6 acupressure on postoperative vomiting in children undergoing outpatient strabismus correction. Br J Anaesth. 1991 Jul;67(1):73-8. doi: 10.1093/bja/67.1.73. PMID 1859764
- [Background] Stein DJ, Birnbach DJ, Danzer BI, Kuroda MM, Grunebaum A, Thys DM. Acupressure versus intravenous metoclopramide to prevent nausea and vomiting during spinal anesthesia for cesarean section. Anesth Analg. 1997 Feb;84(2):342-5. doi: 10.1097/00000539-199702000-00018. PMID 9024025
- [Background] White PF, Issioui T, Hu J, Jones SB, Coleman JE, Waddle JP, Markowitz SD, Coloma M, Macaluso AR, Ing CH. Comparative efficacy of acustimulation (ReliefBand) versus ondansetron (Zofran) in combination with droperidol for preventing nausea and vomiting. Anesthesiology. 2002 Nov;97(5):1075-81. doi: 10.1097/00000542-200211000-00008. PMID 12411789
- [Background] Zarate E, Mingus M, White PF, Chiu JW, Scuderi P, Loskota W, Daneshgari V. The use of transcutaneous acupoint electrical stimulation for preventing nausea and vomiting after laparoscopic surgery. Anesth Analg. 2001 Mar;92(3):629-35. doi: 10.1097/00000539-200103000-00014. PMID 11226090
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupressure Point P6 Stimulator: Acupuncture point P6 stimulation. The device was put on the patients in the operating room prior to administration of the regional anesthesia and was removed after the cesarean section was complete.
Period: Overall Study
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Started | 60 | 60 | 60
Completed | 60 | 60 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator | Total
Number analyzed (Participants) | 60 | 60 | 60 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 60 | 180
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 60 | 180
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 60 | 180

OUTCOME MEASURES:

1. Primary Outcome: Nausea
Description: The investigators will analyze if there is a statistically significant difference between the number of patients that experience nausea at any point during the surgical procedure in each group.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 44 | 14 | 22
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Equivalence — Our null hypothesis is that there is no statistically significant difference between the number of people who experienced nausea in the above 2 groups; p < 0.00001, Chi-squared
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.00005, Chi-squared
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1, Chi-squared

2. Primary Outcome: Vomiting
Description: The investigators will perform objective assessments of whether or not the patients have vomited during the procedure. The investigators will then analyze if there is a statistically significant difference between the number of patients that vomit in each group.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 27 | 10 | 8
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Equivalence — Our null hypothesis is that there is no statistically significant difference between the number of people who experienced vomiting in the above 2 groups; p = 0.001, Chi-squared
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0002, Chi-squared
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.8, Chi-squared

3. Secondary Outcome: Nausea During Stage I (After the Administration of CSE and Until Eversion of the Uterus)
Description: Patients offer their subjective assessments of the level of nausea on a scale of 0-10 (0 = no nausea, 10 = worst nausea ever experienced) during stage I. The investigators will analyze if there is a statistically significant difference between the number of patients that experience nausea in each group at this point. Patients that report nausea (1 or more on our scale) will be recorded as that they have experienced nausea.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 33 | 7 | 14
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.00004, Chi-squared
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0004, Chi-squared
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.09, Chi-squared

4. Secondary Outcome: Nausea During Stage II (After Eversion of the Uterus and Until Replacement of the Uterus)
Description: Patients offer their subjective assessments of the level of nausea on a scale of 0-10 (0 = no nausea, 10 = worst nausea ever experienced) during stage II. The investigators will analyze if there is a statistically significant difference between the number of patients that experience nausea in each group at this point. Patients that report nausea (1 or more on our scale) will be recorded as that they have experienced nausea.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 12 | 6 | 5
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1, Chi-squared
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.07, Chi-squared
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.7, Chi-squared

5. Secondary Outcome: Nausea During Stage III (After Replacement of the Uterus and to the Next 15 Minutes)
Description: Patients offer their subjective assessments of the level of nausea on a scale of 0-10 (0 = no nausea, 10 = worst nausea ever experienced) during stage III. The investigators will analyze if there is a statistically significant difference between the number of patients that experience nausea in each group at this point. Patients that report nausea (1 or more on our scale) will be recorded as that they have experienced nausea.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 16 | 8 | 14
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.7, Chi-squared
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.7, Chi-squared
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.2, Chi-squared

6. Secondary Outcome: Nausea During Stage IV (the Rest of the Time Until Arrival at PACU)
Description: Patients offer their subjective assessments of the level of nausea on a scale of 0-10 (0 = no nausea, 10 = worst nausea ever experienced) during stage IV. The investigators will analyze if there is a statistically significant difference between the number of patients that experience nausea in each group at this point. Patients that report nausea (1 or more on our scale) will be recorded as that they have experienced nausea.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 3 | 4 | 0
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 1, Chi-squared
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.2, Chi-squared
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1, Chi-squared

7. Secondary Outcome: Vomiting During Stage I (After the Administration of CSE and Until Eversion of the Uterus)
Description: The investigators will perform objective assessments of whether or not the patients have vomited during stage I. The investigators will then analyze if there is a statistically significant difference between the number of patients that vomit in each group.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 20 | 5 | 4
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.001, Chi-squared
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0004, Chi-squared
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 1, Chi-squared

8. Secondary Outcome: Vomiting During Stage II (After Eversion of the Uterus and Until Replacement of the Uterus)
Description: The investigators will perform objective assessments of whether or not the patients have vomited during stage II. The investigators will then analyze if there is a statistically significant difference between the number of patients that vomit in each group.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 10 | 1 | 3
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.008, Chi-squared
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.07, Chi-squared
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.6, Chi-squared

9. Secondary Outcome: Vomiting During Stage III (After Replacement of the Uterus and to the Next 15 Minutes)
Description: The investigators will perform objective assessments of whether or not the patients have vomited during stage III. The investigators will then analyze if there is a statistically significant difference between the number of patients that vomit in each group.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 9 | 4 | 6
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.2, Chi-squared
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.5, Chi-squared
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.7, Chi-squared

10. Secondary Outcome: Vomiting During Stage IV (the Rest of the Time Until Arrival at PACU)
Description: The investigators will perform objective assessments of whether or not the patients have vomited during stage IV. The investigators will then analyze if there is a statistically significant difference between the number of patients that vomit in each group.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 0 | 2 | 0
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.5, Chi-squared
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 1, Chi-squared
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.5, Chi-squared

11. Secondary Outcome: Satisfaction of Anti-emetic Treatment
Description: Patients are asked their anti-emetic treatment satisfaction (0 = Not Satisfied, 10 = Extremely Satisfied). Data are expressed as number of parturients who gave a score of 8 or higher.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 49 | 58 | 55
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Superiority — Our null hypothesis is that there is no statistically significant difference between the mean satisfaction level in the above 2 groups; p = 0.02, Fisher Exact
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 11, analysis 1]; p = 0.2, Fisher Exact
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 11, analysis 1]; p = 0.3, Fisher Exact

12. Secondary Outcome: Overall Anesthetic Care Satisfaction
Description: Patients are asked their overall anesthetic care satisfaction (0 = Not Satisfied, 10 = Extremely Satisfied). Data are expressed as number of parturients who gave a score of 8 or higher.
Time Frame: During the surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
Number analyzed (Participants) | 60 | 60 | 60
Participants | 53 | 58 | 56
Statistical Analysis 1: Comparison: Control vs Metoclopramide, Ondansetron; Test type: Equivalence — [test comment as in outcome 11, analysis 1]; p = 0.2, Fisher Exact
Statistical Analysis 2: Comparison: Control vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 11, analysis 1]; p = 0.5, Fisher Exact
Statistical Analysis 3: Comparison: Metoclopramide, Ondansetron vs Acupressure Point P6 Stimulator; Test type: Equivalence — [test comment as in outcome 11, analysis 1]; p = 0.7, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Control | Metoclopramide, Ondansetron | Acupressure Point P6 Stimulator
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes